CLINICAL TRIAL: NCT03727126
Title: Robotic Versus Thoracolaparoscopic Esophagectomy for Carcinoma Esophagus: a Prospective Comparative Study
Brief Title: Robotic Versus Thoracolaparoscopic Esophagectomy for Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMBOT
Record Dates: First submitted 2018-10-27; First posted 2018-11-01 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; Robotic esophagectomy; Laparoscopic esophagectomy; Minimally invasive esophagectomy; Ivor Lewis esophagectomy; McKeown's esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic esophagectomy (Experimental): Esophagectomy performed for esophageal cancer using the da Vinci robotic surgical system
  Interventions: Procedure: Robotic esophagectomy
- Thoracolaparoscopic esophagectomy (Active Comparator): Esophagectomy performed for esophageal cancer using conventional thoracoscopic and laparoscopic techniques
  Interventions: Procedure: Thoracolaparoscopic esophagectomy

INTERVENTIONS:
Procedure: Robotic esophagectomy — Removal of the esophagus and its draining lymph nodes using robotic surgical instruments
  Arms: Robotic esophagectomy
Procedure: Thoracolaparoscopic esophagectomy — Removal of the esophagus and its draining lymph nodes using conventional thoracoscopic and laparoscopic techniques
  Arms: Thoracolaparoscopic esophagectomy

SUMMARY:
Esophageal cancer is a debilitating condition. The treatment involved is complex requiring a combination of chemotherapy and surgery in most cases. Complete removal of the tumor and the adjacent lymph nodes is of utmost importance in improving the survival. Lymph node yield following surgery helps in proper staging of the disease and is an important prognosticating variable. It is hypothesized that the lymph node yield following robotic esophagectomy is higher than that following thoracolaparoscopic esophagectomy. The study aims to compare the short term oncological outcomes following robotic esophagectomy and thoracolaparoscopic esophagectomy for carcinoma esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Resectable esophageal carcinoma, either squamous cell carcinoma or adenocarcinoma in the middle or lower part the esophagus

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) class 4 and above
* Esophagectomy for other non-malignant conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node yield | 7 days after Index Surgery
  Total number of lymph nodes harvested

SECONDARY OUTCOMES:
Surgical margin status | 7 days after Index Surgery
  The proximal, distal and circumferential surgical margins will be assessed by pathological evaluation for the presence of tumor and will be assigned an "R" category as defined by the College of American Pathologists. R0 would indicate no evidence of residual tumor. Presence of microscopic tumor at margins would be designated as R1 whereas the presence of macroscopically visible tumor at margins would be designated as R2.
Complications | Up to 90 days after surgery
  Intraoperative and post operative adverse events assessed by Clavien Dindo classification system
ICU stay | During index admission or within 30 days after surgery
  Duration of stay in ICU following surgery
Hospital stay | During index admission or re admission within 30 days
  Length of stay in hospital following surgery
Mortality | During index admission or within 90 days following surgery
  Death following surgery
Duration of surgery | 1 day after surgery
  Time taken to complete the surgical procedure recorded in minutes
Blood loss | During surgery and up to 24 hours after index surgery
  Amount of blood lost during and within 24 hours of surgery
Conversion rate | 1 day after surgery
  Need for conversion of the procedure to open or other alternate technique

CONTACTS AND LOCATIONS:
Overall Officials: Chinnusamy Palanivelu, MS, MCh, Principal Investigator — GEM Hospital & Research Center; Shankar Balasubramanian, MS, MRCS, Study Director — GEM Hospital & Research Center; Sandeep Sabnis, MS, DNB, Study Director — GEM Hospital & Research Center
Locations (2):
- India (2):
  - GEM Hospital & Research Center, Chennai, Tamil Nadu
  - GEM Hospital & Research Center, Coimbatore, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Undecided